CLINICAL TRIAL: NCT03358147
Title: A Randomized, Double-Blind, Parallel Group, Multi-Center 24-Week Study Comparing the Efficacy and Safety of Three Doses of PT001 to Placebo and Open-label Spiriva® Respimat® in Subjects With Persistent Asthma
Brief Title: Efficacy and Safety of PT001 to Placebo and Open-label Spiriva® Respimat® in Subjects With Persistant Asthma
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Pearl Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PT001102; NCT03547466 (obsolete NCT alias)
Record Dates: First submitted 2017-11-20; First posted 2017-11-30 (Actual); Results first posted 2020-08-12 (Actual); Last update posted 2020-08-12 (Actual); Status verified 2020-08

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Intervention Model Description: Linear repeated measures model
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double Blind vs Placebo, Open Label Spiriva Respimat
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- GP MDI 28.8 μg (Experimental): GP MDI 14.4 μg per actuation taken as 2 inhalations BID
  Interventions: Drug: GP MDI 28.8 μg
- GP MDI 14.4 μg (Experimental): GP MDI 7.2 μg per actuation taken as 2 inhalations BID
  Interventions: Drug: GP MDI 14.4 μg
- GP MDI 7.2 μg (Experimental): GP MDI 3.6 μg per actuation taken as 2 inhalations BID
  Interventions: Drug: GP MDI 7.2 μg
- Placebo MDI (Placebo Comparator): Taken as 2 inhalations BID
  Interventions: Drug: Placebo MDI
- Spiriva Respimat 2.5 μg (Other): Open Label Spiriva Respimat 2.5 μg
  Interventions: Drug: Spiriva Respimat 2.5 μg

INTERVENTIONS:
Drug: GP MDI 28.8 μg — GP MDI (PT001)14.4 μg per actuation taken as 2 inhalations BID
  Other Names: GP
  Arms: GP MDI 28.8 μg
Drug: GP MDI 14.4 μg — GP MDI (PT001) 7.2 μg per actuation taken as 2 inhalations BID
  Other Names: GP
  Arms: GP MDI 14.4 μg
Drug: GP MDI 7.2 μg — GP MDI (PT001) 3.6 μg per actuation taken as 2 inhalations BID
  Other Names: GP
  Arms: GP MDI 7.2 μg
Drug: Placebo MDI — Placebo taken as 2 inhalations BID
  Other Names: Placebo
  Arms: Placebo MDI
Drug: Spiriva Respimat 2.5 μg — Spiriva Respimat 2.5 μg QD (open-label)
  Other Names: Spiriva Respimat
  Arms: Spiriva Respimat 2.5 μg

SUMMARY:
Study Comparing the Efficacy and Safety of PT001 to Placebo and Open-label Spiriva® Respimat® in Subjects With Persistent Asthma

DETAILED DESCRIPTION:
A Randomized, Double-Blind, Parallel Group, Multi-Center 24-Week Study Comparing the Efficacy and Safety of Three Doses of PT001 to Placebo and Open-label Spiriva® Respimat® in Subjects With Persistent Asthma

ELIGIBILITY:
Inclusion Criteria:

* Have a documented history of physician-diagnosed asthma
* Require inhaled asthma maintenance therapy: has been regularly using an ICS/LABA on a stable regimen for at least 4 weeks
* Documented reversibility to albuterol
* A pre-bronchodilator FEV1 >40% and <85% of predicted normal value for subjects 18 to 80 years of age or >40% and <90% of predicted for subjects 12 to <18 years of age
* Demonstrate acceptable spirometry performance
* Willing and, in the opinion of the Investigator, able to adjust current asthma therapy, as required by the protocol
* Compliance: must be willing to remain at the study center as required per protocol to complete all visit assessments

Exclusion Criteria:

* Oral corticosteroid use (any dose) within 4 weeks
* Current smokers, former smokers with >10 pack-years history, or former smokers who stopped smoking <6 months (including all forms of tobacco, e-cigarettes, and marijuana)
* Life-threatening asthma as defined as a history of significant asthma episode(s) requiring intubation associated with hypercapnia, respiratory arrest, hypoxic seizures, or asthma-related syncopal episode(s)
* Completed treatment for lower respiratory infection or asthma exacerbation within 4 weeks
* Hospitalizations for asthma within 3 months
* Historical or current evidence of a clinically significant disease
* Cancer not in complete remission for at least 5 years
* Treatment with investigational study drug (or device) in another clinical study within the last 30 days or 5 half-lives, whichever is longer
* Previously randomized in any PT001 study

Ages: 12 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1077 (Actual)
Dates: Start 2017-12-13 (Actual); Primary Completion 2019-09-12 (Actual); Study Completion 2019-09-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (191):
- United States (191):
  - Research Site, Birmingham, Alabama
  - Research Site, Dothan, Alabama
  - Research Site, Guntersville, Alabama
  - Research Site, Jasper, Alabama
  - Research Site, Scottsboro, Alabama
  - Research Site, Chandler, Arizona
  - Research Site, Flagstaff, Arizona
  - Research Site, Phoenix, Arizona
  - Research Site, Tempe, Arizona
  - Research Site, Tucson, Arizona
  - Research Site, Little Rock, Arkansas
  - Research Site, Anaheim, California
  - Research Site, Bakersfield, California
  - Research Site, Corona, California
  - Research Site, Costa Mesa, California
  - Research Site, El Cajon, California
  - Research Site, Encinitas, California
  - Research Site, Fresno, California
  - Research Site, Fullerton, California
  - Research Site, Gold River, California
  - Research Site, Huntington Beach, California
  - Research Site, Long Beach, California
  - Research Site, Los Angeles, California
  - Research Site, Mission Viejo, California
  - Research Site, Newport Beach, California
  - Research Site, North Hollywood, California
  - Research Site, Northridge, California
  - Research Site, Orange, California
  - Research Site, Palmdale, California
  - Research Site, Poway, California
  - Research Site, Quartz Hill, California
  - Research Site, Rancho Mirage, California
  - Research Site, Riverside, California
  - Research Site, Rolling Hills Estates, California
  - Research Site, Sacramento, California
  - Research Site, San Diego, California
  - Research Site, San Jose, California
  - Research Site, Stockton, California
  - Research Site, Thousand Oaks, California
  - Research Site, Tustin, California
  - Research Site, Westminster, California
  - Research Site, Centennial, Colorado
  - Research Site, Colorado Springs, Colorado
  - Research Site, Lafayette, Colorado
  - Research Site, Wheat Ridge, Colorado
  - Research Site, Hamden, Connecticut
  - Research Site, Aventura, Florida
  - Research Site, Brandon, Florida
  - Research Site, Clearwater, Florida
  - Research Site, Gainesville, Florida
  - Research Site, Hialeah, Florida
  - Research Site, Kissimmee, Florida
  - Research Site, Lake City, Florida
  - Research Site, Loxahatchee Groves, Florida
  - Research Site, Miami, Florida
  - Research Site, Ocala, Florida
  - Research Site, Ocoee, Florida
  - Research Site, Orlando, Florida
  - Research Site, Panama City, Florida
  - Research Site, Pembroke Pines, Florida
  - Research Site, Saint Cloud, Florida
  - Research Site, Tallahassee, Florida
  - Research Site, Tampa, Florida
  - Research Site, Winter Park, Florida
  - Research Site, Adairsville, Georgia
  - Research Site, Albany, Georgia
  - Research Site, Atlanta, Georgia
  - Research Site, Columbus, Georgia
  - Research Site, Dacula, Georgia
  - Research Site, Gainesville, Georgia
  - Research Site, Lawrenceville, Georgia
  - Research Site, Norcross, Georgia
  - Research Site, Rincon, Georgia
  - Research Site, Savannah, Georgia
  - Research Site, Stockbridge, Georgia
  - Research Site, Boise, Idaho
  - Research Site, Meridian, Idaho
  - Research Site, Evergreen Park, Illinois
  - Research Site, O'Fallon, Illinois
  - Research Site, River Forest, Illinois
  - Research Site, Brownsburg, Indiana
  - Research Site, Michigan City, Indiana
  - Research Site, Fort Mitchell, Kentucky
  - Research Site, Crowley, Louisiana
  - Research Site, Shreveport, Louisiana
  - Research Site, Zachary, Louisiana
  - Research Site, Bangor, Maine
  - Research Site, Chevy Chase, Maryland
  - Research Site, White Marsh, Maryland
  - Research Site, Fall River, Massachusetts
  - Research Site, North Dartmouth, Massachusetts
  - Research Site, Ann Arbor, Michigan
  - Research Site, Farmington Hills, Michigan
  - Research Site, Rochester, Michigan
  - Research Site, Troy, Michigan
  - Research Site, Edina, Minnesota
  - Research Site, Fridley, Minnesota
  - Research Site, Minneapolis, Minnesota
  - Research Site, Woodbury, Minnesota
  - Research Site, Chesterfield, Missouri
  - Research Site, Columbia, Missouri
  - Research Site, Saint Charles, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, Bellevue, Nebraska
  - Research Site, Lincoln, Nebraska
  - Research Site, Omaha, Nebraska
  - Research Site, Las Vegas, Nevada
  - Research Site, Reno, Nevada
  - Research Site, Berlin, New Jersey
  - Research Site, Ocean City, New Jersey
  - Research Site, Skillman, New Jersey
  - Research Site, Toms River, New Jersey
  - Research Site, Albuquerque, New Mexico
  - Research Site, Cortland, New York
  - Research Site, New York, New York
  - Research Site, The Bronx, New York
  - Research Site, Watertown, New York
  - Research Site, Burlington, North Carolina
  - Research Site, Charlotte, North Carolina
  - Research Site, Elizabeth City, North Carolina
  - Research Site, Gastonia, North Carolina
  - Research Site, Greensboro, North Carolina
  - Research Site, Hickory, North Carolina
  - Research Site, Huntersville, North Carolina
  - Research Site, Monroe, North Carolina
  - Research Site, Mooresville, North Carolina
  - Research Site, New Bern, North Carolina
  - Research Site, Raleigh, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Fargo, North Dakota
  - Research Site, Cincinnati, Ohio
  - Research Site, Columbus, Ohio
  - Research Site, Dayton, Ohio
  - Research Site, Dublin, Ohio
  - Research Site, Marion, Ohio
  - Research Site, Wooster, Ohio
  - Research Site, Edmond, Oklahoma
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Tulsa, Oklahoma
  - Research Site, Clackamas, Oregon
  - Research Site, Medford, Oregon
  - Research Site, Portland, Oregon
  - Research Site, Monroeville, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Wyomissing, Pennsylvania
  - Research Site, East Providence, Rhode Island
  - Research Site, Warwick, Rhode Island
  - Research Site, Anderson, South Carolina
  - Research Site, Charleston, South Carolina
  - Research Site, Gaffney, South Carolina
  - Research Site, Greenville, South Carolina
  - Research Site, Hodges, South Carolina
  - Research Site, Mt. Pleasant, South Carolina
  - Research Site, Myrtle Beach, South Carolina
  - Research Site, Rock Hill, South Carolina
  - Research Site, Spartanburg, South Carolina
  - Research Site, Union, South Carolina
  - Research Site, Rapid City, South Dakota
  - Research Site, Franklin, Tennessee
  - Research Site, Hendersonville, Tennessee
  - Research Site, Johnson City, Tennessee
  - Research Site, Smyrna, Tennessee
  - Research Site, Amarillo, Texas
  - Research Site, Austin, Texas
  - Research Site, Boerne, Texas
  - Research Site, Carrollton, Texas
  - Research Site, Dallas, Texas
  - Research Site, El Paso, Texas
  - Research Site, Houston, Texas
  - Research Site, Kerrville, Texas
  - Research Site, Killeen, Texas
  - Research Site, Lampasas, Texas
  - Research Site, Live Oak, Texas
  - Research Site, Lufkin, Texas
  - Research Site, Pearland, Texas
  - Research Site, Plano, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Sherman, Texas
  - Research Site, Tomball, Texas
  - Research Site, Waco, Texas
  - Research Site, Murray, Utah
  - Research Site, Salt Lake City, Utah
  - Research Site, South Burlington, Vermont
  - Research Site, Abingdon, Virginia
  - Research Site, Newport News, Virginia
  - Research Site, Richmond, Virginia
  - Research Site, Bellingham, Washington
  - Research Site, Spokane Valley, Washington
  - Research Site, Tacoma, Washington
  - Research Site, Morgantown, West Virginia
  - Research Site, Greenfield, Wisconsin

REFERENCES:
- [Derived] Oba Y, Anwer S, Maduke T, Patel T, Dias S. Effectiveness and tolerability of dual and triple combination inhaler therapies compared with each other and varying doses of inhaled corticosteroids in adolescents and adults with asthma: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2022 Dec 6;12(12):CD013799. doi: 10.1002/14651858.CD013799.pub2. PMID 36472162
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=PT001102&attachmentIdentifier=16b78123-fc13-4fe3-9372-a54985c559e3&fileName=PT001102_SAP_v1.0_2019_08_Redacted_05052020_PDFA.pdf&versionIdentifier=
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=PT001102&attachmentIdentifier=62b683f8-2d58-4502-8424-a59e8275b898&fileName=PT001102_Protocol_Amendment_4_V_5.0_08Mar2019_Redacted_PDFA.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study randomized subjects at 194 sites in the United States from December 2017 to September 2019. The entire study period was scheduled to take up to approximately 26 weeks for each individual subject from the time of screening through the follow up period.
Pre-assignment Details: Subjects were randomized in a 2:2:2:2:1 Scheme to follow 1 of the 5 treatment groups.
Groups:
- GP MDI 28.8 μg: Glycopyrronium Metered Dose Inhalation 28.8 μg
- GP MDI 14.4 μg: Glycopyrronium Metered Dose Inhalation 14.4 μg
- GP MDI 7.2 μg: Glycopyrronium Metered Dose Inhalation 7.2μg
- Placebo MDI: Placebo Metered Dose Inhalation
- Spiriva Respimat 2.5 μg: Spiriva Respimat 2.5 μg
Period: Overall Study
Arm/Group | GP MDI 28.8 μg | GP MDI 14.4 μg | GP MDI 7.2 μg | Placebo MDI | Spiriva Respimat 2.5 μg
Started (6 subjects were excluded due to overlapping IP exposure) | 235 | 240 | 240 | 237 | 119
Completed | 201 | 201 | 206 | 201 | 105
Not Completed | 34 | 39 | 34 | 36 | 14
Not completed — Withdrawal by Subject | 13 | 19 | 16 | 10 | 5
Not completed — Adverse Event | 3 | 9 | 7 | 5 | 2
Not completed — Lost to Follow-up | 4 | 3 | 7 | 6 | 4
Not completed — Major Protocol Deviation | 11 | 3 | 2 | 3 | 1
Not completed — Protocol specified criteria | 2 | 3 | 0 | 3 | 1
Not completed — Physician Decision | 1 | 0 | 1 | 6 | 1
Not completed — Administrative reasons | 0 | 1 | 0 | 3 | 0
Not completed — Lack of Efficacy | 0 | 1 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GP MDI 28.8 μg | GP MDI 14.4 μg | GP MDI 7.2 μg | Placebo MDI | Spiriva Respimat 2.5 μg | Total
Number analyzed (Participants) | 235 | 240 | 240 | 237 | 119 | 1071
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: Safety Population
  Years | 48.4 (15.1) | 47.7 (16.8) | 46.7 (15.5) | 47.1 (16.2) | 49.8 (15.3) | 47.7 (15.8)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Safety Population
  Participants
    Female | 146 | 153 | 151 | 134 | 76 | 660
    Male | 89 | 87 | 89 | 103 | 43 | 411
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Safety Population
  Participants
    Hispanic or Latino | 36 | 61 | 52 | 51 | 21 | 221
    Not Hispanic or Latino | 198 | 179 | 186 | 186 | 98 | 847
    Unknown or Not Reported | 1 | 0 | 2 | 0 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Safety Population
  Participants
    American Indian or Alaska Native | 0 | 1 | 3 | 0 | 1 | 5
    Asian | 6 | 1 | 6 | 2 | 0 | 15
    Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 0 | 0 | 1
    Black or African American | 62 | 68 | 52 | 52 | 25 | 259
    White | 165 | 168 | 177 | 179 | 93 | 782
    More than one race | 0 | 0 | 0 | 0 | 0 | 0
    Unknown or Not Reported | 1 | 2 | 2 | 4 | 0 | 9

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Forced Expiratory Volume in 1 Second (FEV1) Area Under the Curve From 0 to 4 Hours (AUC0-4)
Description: Change from baseline in forced expiratory volume in 1 second (FEV1) area under the curve from 0 to 4 hours (AUC0-4)AUC was normalized for length of follow up (e.g. typically 4 hours).
Time Frame: Week 24
Population: mITT Population
Measure: Least Squares Mean (95% Confidence Interval); unit: Liter
Arm/Group | GP MDI 28.8 μg | GP MDI 14.4 μg | GP MDI 7.2 μg | Placebo MDI | Spiriva Respimat 2.5 μg
Number analyzed (Participants) | 195 | 199 | 205 | 196 | 103
Liter | 0.294 [0.248 to 0.341] | 0.284 [0.238 to 0.331] | 0.308 [0.263 to 0.354] | 0.240 [0.194 to 0.287] | 0.347 [0.282 to 0.412]

2. Secondary Outcome: Change From Baseline in Morning Pre-dose Trough FEV1
Time Frame: Week 24
Population: mITT Population
Measure: Least Squares Mean (95% Confidence Interval); unit: Liter
Arm/Group | GP MDI 28.8 μg | GP MDI 14.4 μg | GP MDI 7.2 μg | Placebo MDI | Spiriva Respimat 2.5 μg
Number analyzed (Participants) | 196 | 199 | 205 | 198 | 102
Liter | 0.142 [0.097 to 0.188] | 0.108 [0.063 to 0.153] | 0.142 [0.098 to 0.187] | 0.129 [0.084 to 0.174] | 0.150 [0.087 to 0.213]

3. Secondary Outcome: Rate of Moderate to Severe Asthma Exacerbations
Description: Rate of moderate to severe Asthma exacerbations (A deterioration of asthma requiring a new or increased dose of ICS for at least 3 days) or severe Asthma exacerbation (Use of systemic corticosteroids (tablets, suspension, or injection) for at least 3 days OR a hospitalization or ER visit because of asthma)
Time Frame: over 24 Weeks (timepoints of 4, 12 & 20 weeks)
Population: mITT Population
Measure: Mean (Standard Error); unit: Events per year
Arm/Group | GP MDI 28.8 μg | GP MDI 14.4 μg | GP MDI 7.2 μg | Placebo MDI | Spiriva Respimat 2.5 μg
Number analyzed (Participants) | 231 | 240 | 240 | 237 | 118
Events per year | 0.43 (0.078) | 0.44 (0.080) | 0.41 (0.076) | 0.55 (0.092) | 0.50 (0.123)

4. Secondary Outcome: Change From Baseline in ACQ-7 (Asthma Control Questionnaire)
Description: ACQ-7: The ACQ, comprising 7 questions, is completed in the clinic and requires subjects to recall their experiences during the previous week (7 days) prior to the study visit. The ACQ-5 measures 5 symptoms (woken at night by symptoms, wake in the morning with symptoms, limitation of daily activities, shortness of breath, and wheeze); the ACQ-6 is these symptom measurements plus daily rescue medication use as recalled by the subject; and the ACQ 7 is the ACQ 6 plus airway caliber as measured by pre-bronchodilator FEV1 percent predicted. Each question is scored on a 7-point scale (generally, 0=no impairment, 6=maximum impairment), the questions are equally weighted, and the ACQ score is the mean of the item responses and therefore ranges from 0 (totally controlled) to 6 (severely uncontrolled.
Time Frame: Week 24
Population: mITT Population
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | GP MDI 28.8 μg | GP MDI 14.4 μg | GP MDI 7.2 μg | Placebo MDI | Spiriva Respimat 2.5 μg
Number analyzed (Participants) | 189 | 189 | 194 | 187 | 93
Scores on a scale | -0.78 [-0.89 to -0.66] | -0.73 [-0.84 to -0.62] | -0.90 [-1.01 to -0.79] | -0.80 [-0.91 to -0.69] | -0.90 [-1.06 to -0.74]

5. Secondary Outcome: Change From Baseline in ACQ-5 (Asthma Control Questionnaire)
Description: ACQ-5:The ACQ-5 measures 5 symptoms (woken at night by symptoms, wake in the morning with symptoms, limitation of daily activities, shortness of breath, and wheeze). Each question is scored on a 7-point scale (generally, 0=no impairment, 6=maximum impairment), the questions are equally weighted, and the ACQ score is the mean of the item responses and therefore ranges from 0 (totally controlled) to 6 (severely uncontrolled).
Time Frame: Week 24
Population: mITT Population
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | GP MDI 28.8 μg | GP MDI 14.4 μg | GP MDI 7.2 μg | Placebo MDI | Spiriva Respimat 2.5 μg
Number analyzed (Participants) | 195 | 198 | 196 | 196 | 98
Scores on a scale | -0.87 [-1.00 to -0.73] | -0.80 [-0.93 to -0.67] | -1.02 [-1.15 to -0.89] | -0.93 [-1.06 to -0.80] | -1.03 [-1.22 to -0.85]

6. Secondary Outcome: Change From Baseline in Asthma Quality of Life Questionnaire for 12 Years and Older (AQLQ +12)
Description: AQLQ +12 - Asthma Quality of Life Questionnaire The AQLQ +12 is a 32-item validated subject-administered questionnaire that was developed to measure the functional problems (physical, emotional, social and occupational) that are most troublesome to adults (≥18 years of age) and adolescents (12 to 17 years of age) with asthma. The 32 questions in the AQLQ +12 are in 4 domains (symptoms, activity limitation, emotional function, and environmental stimuli). All 4 domains contain standard specific questions relating to each domain. Subjects are asked to think about how they have been during the previous 2 weeks. Responses to each of the 32 questions are on a 7-point scale (7=no impairment to 1=severe impairment). The overall AQLQ +12 score is the mean of all 32 responses. Overall scores range from 1=severe impairment to 7=no impairment.
Time Frame: Week 24
Population: mITT Population
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | GP MDI 28.8 μg | GP MDI 14.4 μg | GP MDI 7.2 μg | Placebo MDI | Spiriva Respimat 2.5 μg
Number analyzed (Participants) | 191 | 191 | 191 | 188 | 94
Scores on a scale | 0.89 [0.74 to 1.04] | 0.90 [0.75 to 1.04] | 1.02 [0.87 to 1.16] | 0.96 [0.82 to 1.11] | 1.04 [0.84 to 1.25]

ADVERSE EVENTS:
Time Frame: Serious Adverse events were collected from the time subject signed Informed Consent to the time of the final follow-up telephone call up to approximately 30 weeks. Adverse Events were collected from the time subject was randomized up to approximately 26 weeks.
Description: The safety analysis set was defined as data from all subjects who were randomized to treatment and received any amount of the study treatment
Arm/Group | GP MDI 28.8 μg | GP MDI 14.4 μg | GP MDI 7.2 μg | Placebo MDI | Spiriva Respimat 2.5 μg
All-Cause Mortality (participants affected / at risk) | 0/235 | 0/240 | 0/240 | 0/237 | 0/119
Serious Adverse Events (participants affected / at risk) | 9/235 | 7/240 | 6/240 | 7/237 | 2/119
Other Adverse Events (participants affected / at risk) | 33/235 | 35/240 | 33/240 | 29/237 | 14/119
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GP MDI 28.8 μg (N=235) | GP MDI 14.4 μg (N=240) | GP MDI 7.2 μg (N=240) | Placebo MDI (N=237) | Spiriva Respimat 2.5 μg (N=119)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthritis infective (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Kindey infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Klebsiella bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metapneumovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerbrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Adverse drug reaction (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Non cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adnexal torsion (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Miscarriage of partner (Social circumstances) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Post traumatic pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GP MDI 28.8 μg (N=235) | GP MDI 14.4 μg (N=240) | GP MDI 7.2 μg (N=240) | Placebo MDI (N=237) | Spiriva Respimat 2.5 μg (N=119)
Upper respiratory tract infection (Infections and infestations) | 14 (15) | 14 (14) | 14 (14) | 19 (20) | 6 (7)
Nasopharyngitis (Infections and infestations) | 11 (12) | 15 (19) | 17 (19) | 8 (10) | 2 (2)
Sinusitis (Infections and infestations) | 10 (10) | 7 (8) | 4 (4) | 3 (3) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Drafts of any and all publications or presentations of this study must be submitted at least 30 days prior to submission for publication or presentation to Pearl Therapeutics for review, approval, and to ensure consistency. Pearl Therapeutics has the right to request appropriate modification to correct facts and to represent it's opinions, or the opinions of the publication committee, if these differ with the proposed publication.

DOCUMENTS (2):
  • Study Protocol (2019-03-08): https://cdn.clinicaltrials.gov/large-docs/47/NCT03358147/Prot_000.pdf
  • Statistical Analysis Plan (2019-08-12): https://cdn.clinicaltrials.gov/large-docs/47/NCT03358147/SAP_001.pdf